CLINICAL TRIAL: NCT06488612
Title: Evaluation of the Use of Minced Skin Grafts for Promoting Donor Site Wound Healing After Split-Thickness Skin Grafting: A Prospective Half-side Comparative Study
Brief Title: Evaluation of the Use of Minced Skin Grafts for Promoting Donor Site Wound Healing After Split-Thickness Skin Grafting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelmawla Mohamed, principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med-24-02-09MS
Record Dates: First submitted 2024-03-15; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Traumatic Skin Loss, 2nd and 3rd Degree Burn, Post Tumour Excision - Raw Areas Undergoes Split- Thickness Skin Grafts
Keywords: Split- thickness Skin grafting
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental): A Prospective Half-side Comparative Study, Minced skin grafts will be used on a half of donor site of the same patient
  Interventions: Procedure: Minced skin grafts for donor site

INTERVENTIONS:
Procedure: Minced skin grafts for donor site — After harvesting of STSG using watson's knife and coverage of the recipient site, the excess graft edges will be trimmed and together with any unused graft pieces will be collected in saline filled plate to prevent graft dissecation. Graft pieces will be placed over a rigid surface such as dorsum of a stainless steal jar or pot. Mincing of these small grafts will be done manually using large blade (no. 25) and sharp scissors. The resulting pasty graft mass composed of a large number of minced skin graft particles and a small amount of saline solution will be spread onto one half of the donor site using small dressing forceps.
  Minced skin grafts will not be used on the other half (control side). The entire donor site will be covered with non-adherent absorbable dressing in the form of Vaseline gauze and sterilized cotton-filled dressing followed by elastic compression bandage.

SUMMARY:
Split-thickness skin grafting (STSG) is one of the most commonly performed procedures to achieve wound closure. Most studies are concerned on improving the appearance of scars and shortening the healing time of the recipient sites. However, the management of the donor site usually takes a second consideration.

There is a lack of consensus on the recommended method of donor site management. Donor site morbidity of STSG is usually minimal, but that may not always be the case. Morbidity may include pigmentary abnormalities, prolonged pain and itching, delayed healing, or unfavorable scarring. So, an effort must be taken to find the optimal solution for donor site healing and minimize morbidity.

Small portions of the skin graft left at the end of the procedure or the graft pieces obtained after trimming the edges are usually discarded. There have been some studies demonstrating the benefit of the minced residual skin graft on the donor site, possibly resulting in earlier epithelialization and improving the appearance

DETAILED DESCRIPTION:
The aim of this study is to compare the duration of wound healing, scar quality and cosmetic results of donor sites after split-thickness skin grafting with and without the use of residual graft pieces as minced skin grafts.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing split-thickness skin grafting, between 12 - 60 years of age.

Exclusion Criteria:

* Patients under the age of 12 years or above 60 years.
* Patients with a known tendency for hypertrophic scarring/keloids
* Pregnancy
* Co-morbid factors such as uncontrolled diabetes, ischemic heart disease, renal failure or Collagen vascular disease.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Scar quality | Follow up at 1 month, 3 months, 6 months
  using POSAS scale.
  • Patient Observer Scar Assesment Scale (POSAS) is a validated scale that measures scar quality by evaluating visual, tactile, and sensory characteristics of the scar from two different perspectives: the patient perspective and the surgeons' perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic surgery department, Faculty of medicine, Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Final results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2023 to December 2024